CLINICAL TRIAL: NCT06331273
Title: Impact of "No-touch" Technique on the Outcome of Liver Transplantation for Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Shulan (Hangzhou) Hospital (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Other Study IDs: CT2024-ZJU-OBS3
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Liver Transplantation; No-touch Technique; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HCC patients fulfill Hangzhou criteria and receive LT with "No-touch" technique
  Interventions: Procedure: Liver transplantation with "No-touch" technique
- HCC patients exceed Hangzhou criteria and receive LT with "No-touch" technique
  Interventions: Procedure: Liver transplantation with "No-touch" technique
- HCC patients fulfill Hangzhou criteria and receive LT without "No-touch" technique
- HCC patients exceed Hangzhou criteria and receive LT without"No-touch" technique

INTERVENTIONS:
Procedure: Liver transplantation with "No-touch" technique — The core principle of "no-touch" tumor surgery revolves around avoiding direct contact with the tumor or surrounding tissues as much as possible to minimize the release of cancer cells into the bloodstream or nearby tissues.
  Groups: HCC patients exceed Hangzhou criteria and receive LT with "No-touch" technique; HCC patients fulfill Hangzhou criteria and receive LT with "No-touch" technique

SUMMARY:
The "no-touch" technique has been one of the most important principles of oncological surgery and aimed to prevent seeding and tumor cell dissemination. Previous studies in hepatectomy have shown that no-touch technique surgery can reduce HCC recurrence and improve the survival of patients. However, there is no consensus on whether the no-touch technique in LT for HCC improves the outcomes. This study aims to prospectively include liver transplant patients from multiple transplant centers, collecting their pre-transplant clinical information, post-transplant pathological records and exploring and clarify the correlation between "no-touch" technique and the prognosis of LT patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC based on CT or MRI imaging or needle biopsy confirming a histologic diagnosis of HCC.
2. Patients undergoing deceased donor liver transplantation for the first time.

Exclusion Criteria:

(1) patients who received split LT or simultaneous transplantation, (2) patients who received re-transplantation, (3) patients with macroscopic portal vein tumor thrombosis or other macrovascular invasion, (4) patients with incomplete follow-up or incomplete important parameters records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients who undergoing deceased donor liver transplantation for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free surviavl rate | 2024.4.1-2028.4.1
Overall survival rate | 2024.4.1-2028.4.1
Tumor recurrence rate | 2024.4.1-2028.4.1